CLINICAL TRIAL: NCT01750554
Title: The Influence of a Bupivacaine Digital Nerve Block With the New Continuous Sensor (Rev G) on the Accuracy of SpHb Monitoring.
Brief Title: The Influence of a Bupivacaine Digital Nerve Block Using Rev G.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-00524D
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Patients Undergoing Spine Surgery
Keywords: SpHb; hemoglobin monitoring;bupivacaine digital nerve block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bupivacaine digital nerve block (Experimental): Patients undergoing spine surgery will have a 50/50 chance of being randomized to receive a bupivacaine 0.25% (2 milliliters total) intermediate-acting digital nerve block.
  Interventions: Other: intermediate-acting digital nerve block
- No bupivacaine digital nerve block (No Intervention): Patients undergoing spine surgery will have a 50/50 chance of being randomized to not receive a bupivacaine 0.25% (2 milliliters total) intermediate-acting digital nerve block.

INTERVENTIONS:
Other: intermediate-acting digital nerve block — non-therapeutic Bupivacaine digital nerve block to assess effect on accuracy of diagnostic readings
  Arms: bupivacaine digital nerve block

SUMMARY:
The investigators are proposing to continue investigation to improve the accuracy of the SpHb (continuous hemoglobin monitoring device) by administering an intermediate acting digital nerve block in the finger connected to the SpHb, specifically bupivacaine 0.25% in patients undergoing spine surgery. Bupivacaine is FDA approved and in routine use.

DETAILED DESCRIPTION:
Patients undergoing spine surgery will be randomized to receive (or not) the bupivacaine digital block on the finger attached to the new limited release version of the hemoglobin sensor, RevG. The SpHb reading will be compared to a blood hemoglobin level analyzed in the UCSF Clinical Laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* American Society of Anesthesiologists classification 1, 2 or 3
* Scheduled to undergo spine or hip surgery

Exclusion Criteria:

* Pregnant or nursing
* Patients who in the study investigators clinical judgement would not be suitable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
SpHb (continuous hemoglobin monitor reading) minus tHb (clinical laboratory determined hemoglobin value). | Intermittent (about hourly) hemoglobin checks throughout the surgery.
  Use of a longer acting local anesthetic (bupivacaine) for the digital nerve block will result in SpHb (the non-invasive hemoglobin device) being sufficiently accurate for blood transfusion decisions(≤ 1.0 g/dL difference)
  To assess if using an intermediate-acting digital nerve block will improve the accuracy of the SpHb readings when compared to a blood hemoglobin level analyzed in the UCSF Clinical Laboratories intermittently during the patient's surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States